CLINICAL TRIAL: NCT02084693
Title: Evaluate Survivorship for the Biomet® Comprehensive® Reverse Shoulder Mini Baseplate.
Brief Title: COMPREHENSIVE® REVERSE SHOULDER Mini BasePlate
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: INT.CR.GE1
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-06

CONDITIONS: Rotator Cuff Tear Arthropathy; Osteoporosis; Osteomalacia; Joint; Destruction, Sacroiliac
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Osteoporosis; Osteomalacia | interventions — Comprehensive Metabolic Panel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COMPREHENSIVE: Evaluate Survivorship for the Biomet® Comprehensive® Reverse Shoulder Mini Baseplate.
  Interventions: Device: COMPREHENSIVE

INTERVENTIONS:
Device: COMPREHENSIVE — Comprehensive® Reverse Shoulder products are indicated for use in patients whose shoulder joint has a grossly deficient rotator cuff with severe arthropathy and/or previously failed shoulder joint replacement with a grossly deficient rotator cuff.

SUMMARY:
Evaluate Survivorship for the Biomet® Comprehensive® Reverse Shoulder Mini Baseplate.

DETAILED DESCRIPTION:
The primary objective of this prospective clinical data collection is to evaluate survivorship for the Biomet® Comprehensive® Reverse Shoulder Mini Baseplate. Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes including adverse events, scapular notching, and Constant Score.

All shoulders on which data will be collected are legally marketed and none of the devices are investigational or experimental. FDA has cleared this device via Premarket Notification 510(k) K080642. This data collection effort will document the clinical outcomes of the Comprehensive® Reverse shoulders. The data gathered will be collated and used to provide feedback to designing engineers, support marketing efforts, and answer potential questions from reimbursement agencies.

ELIGIBILITY:
Inclusion Criteria:

Patients / cases to be included in this study shall utilize the following inclusion criteria:

1. Comprehensive Reverse Shoulder Mini Base Plate and Mini Stem in a reverse shoulder configuration.
2. The patient must be anatomically and structurally suited to receive the implants and a functional deltoid muscle is necessary.
3. Grossly deficient rotator cuff with severe arthropathy and/or

   1. Previously failed shoulder joint replacement with a grossly deficient rotator cuff.
   2. Primary total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency, or
   3. Fracture total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency, or
   4. Revision total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency.

Exclusion Criteria:

* The exclusion criteria are the same as the indications stated in the cleared labeling for the device:

Absolute contraindications include infection, sepsis, and osteomyelitis.

Relative contraindications include:

1. Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
2. Osteoporosis.
3. Metabolic disorders which may impair bone formation.
4. Osteomalacia.
5. Distant foci of infections which may spread to the implant site.
6. Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Therefore, patients / cases to be included in this study shall utilize the following inclusion criteria:
  1. The patient must be anatomically and structurally suited to receive the implants and a functional deltoid muscle is necessary.
  2. Grossly deficient rotator cuff with severe arthropathy and/or
     * Previously failed shoulder joint replacement with a grossly deficient rotator cuff.
     * Primary total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency, or
     * Fracture total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency, or
     * Revision total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Survivorship | 1 year
  The primary objective of this prospective clinical data collection is to evaluate survivorship for the Biomet® Comprehensive® Reverse Shoulder Mini Baseplate.

SECONDARY OUTCOMES:
Adverse Events (including dislocation) | 3 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Constant-Murley Shoulder Score | 3 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Radiographic Evaluation (Plain X-ray and CT) | 3 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Scapular Notching | 3 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Constant-Murley Shoulder Score | 1 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Constant-Murley Shoulder Score | 6 Months
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Radiographic Evaluation | 1 year
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes
Radiographic Evaluation | 6 Weeks
  Secondary objectives include validation of implant sizing and hardware options as well as collection of mid-term clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joo Han Oh, Ph.D., Principal Investigator — Bundang Seoul Nat'l University Hospital; Sang Jin Shin, Ph.D., Principal Investigator — Ewha Womans University Mokdong Hospital; Jae Chul Yoo, Ph. D., Principal Investigator — Samsung Medical Center; Yong Girl Rhee, Ph.D., Principal Investigator — Kyung Hee Univ. Hospital; Kyu Chul Noh, Ph.D., Principal Investigator — Gangnam Sacred Heart Hospital
Locations (5):
- South Korea (5):
  - Bunndang Seoul Nat'l Univ. Hospital, Seongnam-si, Seongnam
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gangnam Sacred Heart Hospital, Seoul
  - Kyung Hee Univ Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT02084693/Prot_000.pdf